CLINICAL TRIAL: NCT01963234
Title: Implementing Technology-Assisted Drug Treatment and Relapse Prevention in Federally Qualified Health Centers (FQHCs)
Acronym: Seva
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Dartmouth College (Other); Center for Health Enhancement System Studies (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012-0937; R01DA034279-01 (NIH)
Record Dates: First submitted 2013-10-09; First posted 2013-10-16 (Estimated); Results first posted 2018-07-31 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Substance Use Disorders; HIV
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Seva (Experimental): Up to 100 patients in each of 3 intervention clinics will receive access to the Seva mobile health system for drug use disorders.
  Interventions: Behavioral: Seva

INTERVENTIONS:
Behavioral: Seva — Patients were given access to use Seva. This is a mobile application that uses social and behavioral theories to help support people after alcohol use disorder recovery.

SUMMARY:
Implementing a mobile-phone based system for drug use disorders in primary care settings.

DETAILED DESCRIPTION:
The purpose of the research is to study the impact of a recovery support system called Seva on primary care organizations, where issues such as coordination of care, job satisfaction, and the cost of adopting and operating new technologies are critical. The study will also investigate how to best implement this kind of technology into health care delivery systems that care for people diagnosed with substance abuse.

ELIGIBILITY:
Inclusion Criteria:

Patient subjects must be 1) age 18 or older 2) meet criteria for Substance Use Disorder (SUD) according to the clinic. Clinician subjects referring patients will ensure that patients: 3) have no current psychotic disorder severe enough to prevent participation, 4) have no acute medical problem requiring immediate inpatient treatment, 5) are willing to use Seva, and 6) can understand and sign a consent form in English.

Clinician subjects include MDs, behavioral health providers, nurses and management staff from the clinics' primary care and behavioral health departments. Clinician must have an interest in the research objectives.

Exclusion Criteria:

* Failure to meet inclusion criteria above will exclude patients and clinicians from participating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 439 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Partnership Health Center, Missoula, Montana
  - Institute for Family Health, The Bronx, New York
  - UW Health Access Clinic, Madison, Wisconsin

REFERENCES:
- [Derived] Quanbeck A. Using Stakeholder Values to Promote Implementation of an Evidence-Based Mobile Health Intervention for Addiction Treatment in Primary Care Settings. JMIR Mhealth Uhealth. 2019 Jun 7;7(6):e13301. doi: 10.2196/13301. PMID 31237841
- [Derived] Mares ML, Gustafson DH, Glass JE, Quanbeck A, McDowell H, McTavish F, Atwood AK, Marsch LA, Thomas C, Shah D, Brown R, Isham A, Nealon MJ, Ward V. Implementing an mHealth system for substance use disorders in primary care: a mixed methods study of clinicians' initial expectations and first year experiences. BMC Med Inform Decis Mak. 2016 Sep 29;16(1):126. doi: 10.1186/s12911-016-0365-5. PMID 27687632
- [Derived] Quanbeck AR, Gustafson DH, Marsch LA, McTavish F, Brown RT, Mares ML, Johnson R, Glass JE, Atwood AK, McDowell H. Integrating addiction treatment into primary care using mobile health technology: protocol for an implementation research study. Implement Sci. 2014 May 29;9:65. doi: 10.1186/1748-5908-9-65. PMID 24884976

RESULTS

PARTICIPANT FLOW:
Groups:
- Seva - Patients: Up to 100 patients in each of 3 intervention clinics will receive access to the Seva mobile health system for drug use disorders.
- Seva - Clinicians: We will analyze data of clinicians who use Seva (e.g. clinical adoption).
Period: Overall Study
Arm/Group | Seva - Patients | Seva - Clinicians
Started | 268 | 171
Completed | 207 | 171
Not Completed | 61 | 0

BASELINE CHARACTERISTICS:
Groups:
- Seva - Madison Site; Seva - Missoula; Seva - Bronx: Patients will receive access to the Seva mobile health system for drug use disorders. Data on clinician participants were not collected due to the focus of the study being the patient.
- Total: Total of all reporting groups
Arm/Group | Seva - Madison Site | Seva - Missoula | Seva - Bronx | Total
Number analyzed (Participants) | 97 | 100 | 71 | 268
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 97 | 100 | 71 | 268
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 40 | 35 | 127
  Male | 45 | 60 | 36 | 141
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 35 | 38
  Not Hispanic or Latino | 96 | 98 | 36 | 230
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 8 | 1 | 13
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 30 | 2 | 35 | 67
  White | 63 | 89 | 24 | 176
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 11 | 11
Region of Enrollment [Number; unit: participants]
  United States | 97 | 100 | 71 | 268
Insured by medicare [Count of Participants; unit: Participants] | 8 | 12 | 8 | 28
Insured by medicaid [Count of Participants; unit: Participants] | 55 | 23 | 33 | 111
Insured by private/other [Count of Participants; unit: Participants] | 18 | 19 | 20 | 57
Not insured [Count of Participants; unit: Participants] | 16 | 46 | 10 | 72
Patient-centered medical home (PCMH) designation [Number; unit: Level] — Three levels of recognition exist, based on practice sites meeting six standards. Level three clinics have the best adherence to the standards. Those standards include team-based care and practice organization, knowing and managing patients, patient-centered access and continuity, care management and support, care coordination and care transitions, and performance measurement and quality improvement.
  Level | 3 | 3 | 3 | NA — Site specific.
Patients enrolled in Seva [Count of Participants; unit: Participants] | 97 | 100 | 71 | 268
Any drinking days [Mean (Standard Deviation); unit: days] — within the last 30 days. Population: Participants dropped out over the duration of the study. Data for each specific clinic was not collected and analyzed. Data was collected and analyzed at the total level for all three clinics.
  days
    number analyzed (Participants) | 72 | 74 | 61 | 207
    (all) | NA (NA) — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA (NA) — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA (NA) — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | 2.53 (6.01)
Risky drinking days [Mean (Standard Deviation); unit: days] — within the last 30 days. Population: Participants dropped out over the duration of the study. Data for each specific clinic was not collected and analyzed. Data was collected and analyzed at the total level for all three clinics.
  days
    number analyzed (Participants) | 72 | 74 | 61 | 207
    (all) | NA (NA) — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA (NA) — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA (NA) — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | 1.25 (3.78)
Illicit drug-use days [Mean (Standard Deviation); unit: days] — within the last 30 days. Population: Participants dropped out over the duration of the study. Data for each specific clinic was not collected and analyzed. Data was collected and analyzed at the total level for all three clinics.
  days
    number analyzed (Participants) | 72 | 74 | 60 | 206
    (all) | NA (NA) — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA (NA) — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA (NA) — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | 3.22 (7.57)
Overall quality of life (QoL) [Mean (Standard Deviation); unit: score on a scale] — Higher scores on the scale indicate higher quality of life. Scale ranges from 8 to 40. It includes mental and physical health sub scale values. These values are summed Population: Participants dropped out over the duration of the study. Data for each specific clinic was not collected and analyzed. Data was collected and analyzed at the total level for all three clinics.
  score on a scale
    number analyzed (Participants) | 71 | 72 | 59 | 202
    (all) | NA (NA) — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA (NA) — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA (NA) — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | 28.47 (6.46)
Physical subscale Quality of Life [Mean (Standard Deviation); unit: score on a scale] — Higher scores on the scale indicate higher quality of life. It includes 4 items on overall physical health, physical function, pain, and fatigue that each has a scale ranging from 1 to 5. These values are summed. Scale ranges from 4 to 20. Population: Participants dropped out over the duration of the study. Data for each specific clinic was not collected and analyzed. Data was collected and analyzed at the total level for all three clinics.
  score on a scale
    number analyzed (Participants) | 72 | 74 | 60 | 206
    (all) | NA (NA) — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA (NA) — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA (NA) — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | 13.2 (3.01)
Mental subscale Quality of Life [Mean (Standard Deviation); unit: score on a scale] — Higher scores on the scale indicate higher quality of life. There are 4 questions that have scales that range from values of 1 to 5. These values are summed to give the score for the mental subscale quality of life. Scale ranges from 4 to 20. Population: Participants dropped out of the study over the duration.
  score on a scale
    number analyzed (Participants) | 71 | 73 | 60 | 204
    (all) | NA (NA) — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA (NA) — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA (NA) — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | 9.75 (2.99)
Number of hospitalizations [Mean (Standard Deviation); unit: hospitalizations] — Within the last 6 months. Population: Participants dropped out of the study over the duration.
  hospitalizations
    number analyzed (Participants) | 72 | 74 | 61 | 207
    (all) | NA (NA) — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA (NA) — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA (NA) — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | 0.43 (1.03)
Number of ER visits [Mean (Standard Deviation); unit: ER visits] — within the past 6 months. Population: Participants dropped out over the duration of the study.
  ER visits
    number analyzed (Participants) | 72 | 74 | 61 | 207
    (all) | NA (NA) — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA (NA) — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA (NA) — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | 1.10 (2.79)
Any drink [Number; unit: participants] — within the last 30 days. Population: Participants dropped out over the duration of the study.
  participants
    number analyzed (Participants) | 72 | 74 | 61 | 207
    (all) | NA — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | 64
Illicit drug use [Number; unit: participants] — within the last 30 days. Population: Participants dropped out of the study over time.
  participants
    number analyzed (Participants) | 72 | 74 | 60 | 206
    (all) | NA — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | 63
Any drink or drug [Number; unit: participants] — within the last 30 days. Population: Participants dropped out of the study over time.
  participants
    number analyzed (Participants) | 72 | 74 | 60 | 206
    (all) | NA — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | 97
Currently receive other addiction treatment [Number; unit: participants] — within the last 6 months. Population: Participants dropped out over time.
  participants
    number analyzed (Participants) | 72 | 74 | 61 | 207
    (all) | NA — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | 89
HIV risky behavior [Number; unit: participants] — within the last 6 months. Population: Participants dropped out over time.
  participants
    number analyzed (Participants) | 72 | 74 | 61 | 207
    (all) | NA — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | 76
HIV testing [Number; unit: participants] — within the past 6 months. Population: Participants dropped out over time.
  participants
    number analyzed (Participants) | 72 | 74 | 60 | 206
    (all) | NA — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | NA — Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others. | 81
Drug of choice is alcohol [Count of Participants; unit: Participants] | 34 | 44 | 27 | 105
Drug of choice is Opiates [Count of Participants; unit: Participants] | 31 | 14 | 8 | 53
Drug of choice is crack cocaine [Count of Participants; unit: Participants] | 9 | 3 | 11 | 23
Drug of choice is marijuana [Count of Participants; unit: Participants] | 1 | 4 | 16 | 21
Drug of choice is methamphetamine [Count of Participants; unit: Participants] | 0 | 15 | 1 | 16
Drug of choice is multiple drugs [Count of Participants; unit: Participants] | 22 | 20 | 8 | 50

OUTCOME MEASURES:

1. Primary Outcome: Implementation Status
Description: The number of implementation milestones completed
Time Frame: up to 3 years
Population: These are milestones achieved for each site.
Measure: Number; unit: milestones
Units Other Than Participants: Milestones
Groups:
- Seva - Madison Site; Seva - Missoula; Seva - Bronx: We identified 12 milestones for to meet for each site.
Arm/Group | Seva - Madison Site | Seva - Missoula | Seva - Bronx
Number analyzed (Participants) | 72 | 74 | 61
Number analyzed (Milestones) | 12 | 12 | 12
milestones | 12 | 12 | 12

2. Primary Outcome: Any Drinking Days in Last 30 Days
Time Frame: 6 months
Population: Measure analyzed as a total among all three clinics. We told clinics that we would not report at the site level. We believed that it could reflect poorly on the organization if a site appeared poorly with regard to outcomes in relation to others.
Measure: Mean (Standard Deviation); unit: days
Groups:
- Seva: Patients in each of 3 intervention clinics who received access to the Seva mobile health system for drug use disorders.
Arm/Group | Seva
Number analyzed (Participants) | 207
days | 1.67 (4.69)

3. Primary Outcome: Risky Drinking Days in the Last 30 Days
Description: Analysis for measure was done for the total of all three sites combined.
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Seva
Number analyzed (Participants) | 207
days | 0.70 (2.58)

4. Primary Outcome: Illicit Drug-use Within the Last 30 Days
Description: Analysis for measure was done for the total of all three sites combined.
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Seva
Number analyzed (Participants) | 206
days | 2.14 (6.55)

5. Primary Outcome: Overall Quality of Life
Description: Analysis for measure was done for the total of all three sites combined. Higher values represent better quality of life. Value was calculated by adding the mental and physical subscale values. Values could range from 8 to 40.
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Seva
Number analyzed (Participants) | 202
score on a scale | 30.03 (7.11)

6. Primary Outcome: Physical Subscale Quality of Life
Description: Analysis for measure was done for the total of all three sites combined. Higher values represent better quality of life. This scare consisted of 4 questions that had scales ranging from 1 to 5. The scores were summed and values could range from 4 to 20.
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Seva
Number analyzed (Participants) | 206
score on a scale | 13.48 (3.11)

7. Primary Outcome: Mental Subscale Quality of Life
Description: Analysis for measure was done for the total of all three sites combined. Higher values represent better quality of life. This consisted of 4 questions that had scaled ranging from 1 to 5. The scores of the scales were summed and values could range from 4 to 20.
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Seva
Number analyzed (Participants) | 204
score on a scale | 10.77 (3.50)

8. Primary Outcome: Patient Had Any Drink Within the Last 30 Days
Description: Analysis for measure was done for the total of all three sites combined.
Time Frame: 6 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Seva
Number analyzed (Participants) | 207
Participants | 51

9. Primary Outcome: Patient Had Illicit Drug Use Within the Last 30 Days
Description: Analysis for measure was done for the total of all three sites combined.
Time Frame: 6 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Seva
Number analyzed (Participants) | 206
Participants | 36

10. Primary Outcome: Patient Had Any Drink or Drug Use Within the Last 30 Days
Description: Analysis for measure was done for the total of all three sites combined.
Time Frame: 6 months
Population: Overall number of participants analyzed because data was self reported and patients were allowed to not answer questions if they chose.
Measure: Count of Participants; unit: Participants
Arm/Group | Seva
Number analyzed (Participants) | 204
Participants | 69

11. Primary Outcome: Patients, Within the Last 6 Months Have Received Other Addiction Treatment
Description: Analysis for measure was done for the total of all three sites combined.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Seva
Number analyzed (Participants) | 207
Participants | 78

12. Primary Outcome: Patients Partook in HIV Risky Behavior in the Last 6 Months
Description: Analysis for measure was done for the total of all three sites combined.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Seva
Number analyzed (Participants) | 207
Participants | 65

13. Primary Outcome: Patients Partook in HIV Testing in the Last 6 Months
Description: Analysis for measure was done for the total of all three sites combined.
Time Frame: 6 months
Population: Overall number of participants analyzed is lower because data is self reported and patients could chose not to answer some questions.
Measure: Count of Participants; unit: Participants
Arm/Group | Seva
Number analyzed (Participants) | 206
Participants | 116

14. Secondary Outcome: Number of Patients Using System
Description: Analysis for measure was done for the total of all three sites combined.
Time Frame: up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | Seva
Number analyzed (Participants) | 268
Participants | 268

15. Secondary Outcome: Clinical Adoption
Description: We analyzed computerized system log files to produce patterns of system adoption of the staff.
Time Frame: up to 3 years
Population: This is the number of primary care clinical staff at the 3 sites who adopted using Seva.
Measure: Count of Participants; unit: Participants
Groups:
- Seva - Clinicians: This is the number of clinicians who work within clinics where Seva was implemented.
Arm/Group | Seva - Clinicians
Number analyzed (Participants) | 171
Participants | 171

16. Secondary Outcome: Total Costs for Clinic
Description: This includes the clinic operating costs and clinic implementation costs of the intervention.
Time Frame: 6 months
Population: This outcome measure was analyzed at the clinic level. Thus, NA is indicated for "Overall number of participants analyzed."
Measure: Number; unit: US dollars
Units Other Than Participants: clinic
Groups:
- Seva - Madison Site; Seva - Missoula; Seva - Bronx: Patients will receive access to the Seva mobile health system for drug use disorders.
Arm/Group | Seva - Madison Site | Seva - Missoula | Seva - Bronx
Number analyzed (Participants) | NA | NA | NA
Number analyzed (clinic) | 1 | 1 | 1
US dollars | 123584 | 140495 | 111298

ADVERSE EVENTS:
Time Frame: Up to 1 year.
Groups:
- Seva - Patients: Patients will receive access to the Seva mobile health system for drug use disorders.
- Seva - Clinicians: Clinicians who worked at Seva sites were also monitored for Adverse events.
Arm/Group | Seva - Patients | Seva - Clinicians
All-Cause Mortality (participants affected / at risk) | 3/268 | 0/171
Serious Adverse Events (participants affected / at risk) | 3/268 | 0/171
Other Adverse Events (participants affected / at risk) | 0/268 | 0/171
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Seva - Patients (N=268) | Seva - Clinicians (N=171)
Death (General disorders) | 2 (2) | 0 (0) — These deaths were non-study related.
Death (General disorders) | 1 (1) | 0 (0) — This was a non-study related death. This participant died of Chronic Obstructive Pulmonary Disease and emphysema.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-05-05): https://cdn.clinicaltrials.gov/large-docs/34/NCT01963234/Prot_SAP_000.pdf